CLINICAL TRIAL: NCT04157387
Title: Effect of Cyriax Inferior Capsule Stretching in Idiopathic Adhesive Capsulitis
Brief Title: Cyriax Inferior Capsule Stretching in Idiopathic Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Ramsha Tariq
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Cyriax Manual Therapy; Stretching
MeSH Terms: conditions — Bursitis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyriax inferior capsular stretching + Manual Therapy (Experimental): Cyriax inferior capsular stretching
  + Electrotherapy Manual therapy : Kaltenborn grade 1 and 2 Mobilization
  Active ROM exercises :
  Home plan include :, wall walking exercises, pendulum exercises ,towel stretch exercises, Cross Body Adduction
  Interventions: Other: Cyriax inferior capsular stretching + Manual Therapy
- Manual Therapy (Active Comparator): Analgesic short-wave diathermy Manual Therapy: Kalternbon grade 1 and 2 Mobilization :, Home plan include :, wall walking exercises, pendulum exercises ,towel stretch exercises, Cross Body Adduction.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Cyriax inferior capsular stretching + Manual Therapy — Electro-therapy 10mins Manual therapy : Kalternbon grade 1 and 2 Mobilization : Inferior glide (10x3), posterior glide, (10 reps x 3 sets), anterior glide (10 reps x 3 sets), Active ROM exercises : 10 reps x 3 sets Home plan include :, wall walking exercises, pendulum exercises ,towel stretch exercises, Cross Body Adduction (10reps x 2 sets ,each) Cyriax inferior capsular stretching
  Arms: Cyriax inferior capsular stretching + Manual Therapy
Other: Manual therapy — Before starting capsule stretching technique, Analgesic short-wave diathermy may be given for 10 minutes.
  Kalternbon grade 1 and 2 Mobilization : Inferior glide (10x3), posterior glide, (10 reps x 3 sets), anterior glide (10 reps x 3 sets), Home plan include :, wall walking exercises, pendulum exercises ,towel stretch exercises, Cross Body Adduction (10reps x 2 sets ,each)
  Arms: Manual Therapy

SUMMARY:
The objective of study is to find out the effectiveness of cyriax capsular stretching in idiopathic adhesive capsulitis and to find out the combined effect of capsular stretching's, mobilization and conservative treatment on pain and Range of Motion (ROM) in idiopathic adhesive capsulitis.

DETAILED DESCRIPTION:
This Randomized study was carried out at Pakistan Railway Hospital Rawalpindi. A total of 28 patients were screened out as per inclusion criteria and randomly placed into two groups A and B through lottery method. The Visual Analogue scale, Shoulder Pain and Disability Index, and Range of Motion of shoulder joint were used as outcome measures. All the patients were assessed at baseline before intervention and at the completion of 3weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Adhesive capsulitis phase 1 and phase 2
* Follow capsular pattern ( ER > Abduction> IR)

Exclusion Criteria:

* Adhesive capsulitis phase 3
* Any intrinsic etiology i.e. rheumatoid arthritis,
* infection,
* gout,
* haemarthrosis or
* tumor or Arthritis in stage III or in stage II with a spastic end-feel

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Goniometer | 3rd week
  Changes from the baseline, Measure the available range of motion or the position of the shoulder joint - typically this is a measure of passive motion like External Rotation, External Rotation and Internal Rotation.
Visual Analogue Scale (VAS) | 3rd Week
  Changes from the baseline, Normative values are not presented so by using a ruler , the score is calculated by measure the distance on 10cm line between the "no pain" point and the patient's mark, provide a range of score from 0-100. A higher score indicates greater pain intensity.
Shoulder pain and disability index (SPADI) | 3rd week
  Changes from the Baseline, SPADI is a self-administered questionnaire that aims to measure pain and disability associated with shoulder disease. It consists of two dimensions, one for pain and second for functional activities.
  The pain element consists of five questions regarding severity of pain and to measure the degree of severity that an individual faced during various activities of daily life that involve upper extremity use. There are eight questions.
  Each subscale is summed up and a total SPADI score is expressed as a percentage.Total pain score : --/50 ×100 = %, Total disability score: --/80 × 100 = %, Total SPADI score: --/130 × 100 = %.
  A score of 0 indicates best 100 indicates worst. A higher score shows more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No